CLINICAL TRIAL: NCT04414566
Title: Induction Chemotherapy Plus Radiotherapy Alone Versus Induction Chemotherapy Plus Concurrent Chemoradiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma: a Phase 3, Multicentre, Randomised Controlled Trial
Brief Title: Induction Chemotherapy Plus Radiotherapy Alone in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Principal Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020HXFH037
Record Dates: First submitted 2020-05-24; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Induction Chemotherapy; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Docetaxel; Fluorouracil; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IC plus RT (Experimental): Patients receive GP(gemcitabine+cisplatin) or TPF(docetaxel+cisplatin+fluorouracil) every three weeks for three cycles before the radiotherapy, and then receive radical radiotherapy and cisplatin (100mg/m^2) every three weeks for three cycles during radiotherapy.
  Interventions: Drug: gemcitabine and cisplatin; docetaxel, cisplatin and fluorouracil; Radiation: IMRT
- IC plus CCRT (Active Comparator): Patients receive GP(gemcitabine+cisplatin) or TPF(docetaxel+cisplatin+fluorouracil) every three weeks for three cycles before the radiotherapy, and then receive radical radiotherapy.
  Interventions: Drug: gemcitabine and cisplatin; docetaxel, cisplatin and fluorouracil; Radiation: IMRT and concurrent cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin; docetaxel, cisplatin and fluorouracil — Patients receive GP gemcitabine (1000 mg/m^2 d1,8) and cisplatin (80mg/m^2 d1) or TPF docetaxel (60mg/m^2 on day 1), cisplatin (60mg/m^2 on day 1) and fluorouracil (600mg/m^2 on Days 1 to 5) every three weeks for three cycles before the radiotherapy.
  Other Names: GP;TPF
Radiation: IMRT — Intensity modulated-radiotherapy (IMRT) is given as 2.0 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor.
  Arms: IC plus RT
Radiation: IMRT and concurrent cisplatin — Intensity modulated-radiotherapy (IMRT) is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor, concurrently with cisplatin 100 mg/m^2 every 3 weeks for 3 cycles.
  Arms: IC plus CCRT

SUMMARY:
The purpose of this study is to compare induction chemotherapy (TPF or GP) plus radiotherapy alone with induction chemotherapy plus concurrent chemoradiotherapy in patients with locoregionally advanced nasopharyngeal carcinoma (LA-NPC).

ELIGIBILITY:
Inclusion Criteria:

* Newly pathologically confirmed as non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated, ie WHO type II or III).
* Age ≥ 18 and ≤ 65 years old.
* Tumor staged as III/IVa (according to the 8th AJCC edition).
* No evidence of distant metastasis (M0).
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: White blood cells (WBC) ≥ 4 × 10^9/L, hemoglobin (HGB) ≥ 90 g/L, platelets (PLT) ≥ 100 × 10^9/L (or within the normal range of the laboratory)
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min.
* Written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age > 65 or < 18.
* Treatment with palliative intent.
* Previous history of malignant tumors, well-treated basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ outer.
* Pregnancy or lactation.
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume), chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any other serious diseases, which may bring greater risk or affect the compliance of the test, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-year
  Disease-free survival rate is calculated from the date of randomization to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Locoregional recurrence-free survival | 3-year
  Locoregional recurrence-free survival is calculated from randomization to the first locoregional recurrence.
Distant metastasis-free survival | 3-year
  Distant metastasis-free survival is calculated from randomization to the first remote metastases.
Objective response rates after treatments | At the end of Cycle 3 of induction chemotherapy (each cycle is 21 days) and 16 weeks after completion of radiotherapy
Number of participants with adverse events | Every week during treatment, up to 4 weeks after treatment.
  Incidence of acute toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- Xingchen Peng, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No